CLINICAL TRIAL: NCT01431326
Title: Pharmacokinetics of Understudied Drugs Administered to Children Per Standard of Care
Acronym: PTN_POPS
Status: Completed | Type: Observational
Sponsor: Daniel Benjamin (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Daniel Benjamin, Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Other Study IDs: Pro00029638; IND 113645 (Other: FDA); IND 114369 (Other: FDA); IND 114531 (Other: FDA); IND 118358 (Other: FDA); HHSN20100006 (Other Grant/Funding Number: NICHD); HHSN27500020 (Other Grant/Funding Number: NICHD); HHSN27500027 (Other Grant/Funding Number: NICHD); HHSN27500043 (Other Grant/Funding Number: NICHD); HHSN27500049 (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2011-08-17; First posted 2011-09-09 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Adenovirus; Anesthesia; Anxiety; Anxiolysis; Autism; Autistic Disorder; Bacterial Meningitis; Bacterial Septicemia; Benzodiazepine; Bipolar Disorder; Bone and Joint Infections; Central Nervous System Infections; Convulsions; Cytomegalovirus Retinitis; Early-onset Schizophrenia Spectrum Disorders; Epilepsy; General Anesthesia; Gynecologic Infections; Herpes Simplex Virus; Infantile Hemangioma; Infection; Inflammation; Inflammatory Conditions; Intra-abdominal Infections; Lower Respiratory Tract Infections; Migraines; Pain; Pneumonia; Schizophrenia; Sedation; Seizures; Skeletal Muscle Spasms; Skin and Skin-structure Infections; Treatment-resistant Schizophrenia; Urinary Tract Infections; Withdrawal; Sepsis; Gram-negative Infection; Bradycardia; Cardiac Arrest; Cardiac Arrhythmia; Staphylococcal Infections; Nosocomial Pneumonia; Neuromuscular Blockade; Methicillin Resistant Staphylococcus Aureus; Endocarditis; Neutropenia; Headache; Fibrinolytic Bleeding; Pulmonary Arterial Hypertension; CMV Retinitis; Hypertension; Chronic Kidney Diseases; Hyperaldosteronism; Hypokalemia; Heart Failure; Hemophilia; Heavy Menstrual Bleeding; Insomnia
Keywords: adenovirus; anaesthetic; anesthesia; anticoagulant; anti-epileptic; anti-inflammatory; antimicrobial; anti-psychotic; antiviral; anxiety; anxiolysis; anxiolytic; autism; autistic disorder; benzodiazepine; bipolar disorder; convulsions; epilepsy; headaches; herpes simplex virus; herpes simplex virus (HSV); hypertension; infantile hemangioma; infection; inflammation; influenza; lower respiratory tract infection (LRTI); meningitis; migraines; muscle spasms; pain; pneumonia; prophylaxis; retinitis; schizophrenia; sedation; sedative; seizures; septicemia; swelling; urinary tract infection; urinary tract infection (UTI); withdrawal; empiric therapy; staphylococci; Fibrinolytic Bleeding; pulmonary arterial hypertension; CMV retinitis; control of serum phosphorus; Hyperaldosteronism; hypokalemia; heart failure; hemophilia; Heavy Menstrual Bleeding; insomnia
MeSH Terms: conditions — Adenoviridae Infections; Anxiety Disorders; Autistic Disorder; Meningitis, Bacterial; Bipolar Disorder; Central Nervous System Infections; Seizures; Cytomegalovirus Retinitis; Epilepsy; Herpes Simplex; Hemangioma, Capillary; Infections; Inflammation; Intraabdominal Infections; Migraine Disorders; Pain; Pneumonia; Schizophrenia; Schizophrenia, Treatment-Resistant; Urinary Tract Infections; Sepsis; Bradycardia; Heart Arrest; Arrhythmias, Cardiac; Staphylococcal Infections; Healthcare-Associated Pneumonia; Endocarditis; Neutropenia; Headache; Pulmonary Arterial Hypertension; Hypertension; Renal Insufficiency, Chronic; Hyperaldosteronism; Hypokalemia; Heart Failure; Hemophilia A; Menorrhagia; Sleep Initiation and Maintenance Disorders; Influenza, Human; Meningitis; Spasm; Retinitis | interventions — Cidofovir; Ciprofloxacin; Methylprednisolone; Tobramycin; Alfentanil; Clozapine; Haloperidol; Lurasidone Hydrochloride; Molindone; Pentobarbital; Warfarin; ziprasidone; Amikacin; Cefepime; Nafcillin; Piperacillin, Tazobactam Drug Combination; Rocuronium; Vecuronium Bromide; Vancomycin; Aminocaproic Acid; Bosentan; Fosfomycin; Labetalol; Nifedipine; Oxycodone; Sevelamer; Spironolactone; Tranexamic Acid; Zolpidem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: The POPS study is collecting PK data on children prescribed the following drugs of interest per standard of care:
  Other Names: cidofovir; ciprofloxacin; methylprednisolone; tobramycin; alfentanil; clozapine; haloperidol; lurasidone; molindone; pentobarbital; warfarin (oral); ziprasidone; amikacin; cefepime; nafcillin; piperacillin-tazobactam; rocuronium; vecuronium; vancomycin; aminocaproic acid; bosentan; fosfomycin; labetalol; nifedipine; oxycodone; sevelamer carbonate; spironolactone; tranexamic acid; zolpidem

SUMMARY:
Understudied drugs will be administered to children per standard of care as prescribed by their treating caregiver and only biological sample collection during the time of drug administration will be involved. A total of approximately 7000 children aged <21 years who are receiving these drugs for standard of care will be enrolled and will be followed for up a maximum of 90 days. The goal of this study is to characterize the pharmacokinetics of understudied drugs for which specific dosing recommendations and safety data are lacking. The prescribing of drugs to children will not be part of this protocol. Taking advantage of procedures done as part of routine medical care (i.e. blood draws) this study will serve as a tool to better understand drug exposure in children receiving these drugs per standard of care. The data collected through this initiative will also provide valuable pharmacokinetic and dosing information of drugs in different pediatric age groups as well as special pediatric populations (i.e. obese).

DETAILED DESCRIPTION:
The purpose of this study is to characterize the PK ( Pharmacokinetics) of understudied drugs administered to children per standard of care as prescribed by their treating caregiver. This will be accomplished by the collection of biological samples during the time of drug administration per standard of care as prescribed by the caregiver. The prescribing of drugs to children will not be part of this protocol.

Aim #1: Evaluate the PK of understudied drugs currently being administered to children.

Hypothesis #1: The PK of understudied drugs in children will differ from adults and within children according to pediatric age groups or special population.

Aim #2: Explore the pharmacodynamics (PD) of understudied drugs currently being administered to children.

Hypothesis #2: The PD of targeted drugs in children will differ from adults.

Aim #3: Evaluate the influence of genetic factors, metabolic and protein profiles on therapeutic exposure.

Hypothesis #3: Genetic polymorphisms in drug metabolizing enzymes and metabolic and proteomic profiles will impact drug exposure in children.

ELIGIBILITY:
Inclusion Criteria:

* 1) Children (< 21 years of age) who are receiving understudied drugs of interest per standard of care as prescribed by their treating caregiver

Exclusion Criteria:

* 1) Failure to obtain consent/assent (as indicated)
* 2) Known pregnancy as determined via interview or testing if available.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (<21 years of age) receiving drugs per standard of care as prescribed by treating caregiver
Sampling Method: Non-Probability Sample
Enrollment: 3520 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic outcomes for understudied drugs in children | Data will be collected throughout the hospital or outpatient stay up to 90 days
  As appropriate for each study drug, the following additional PK parameters will be estimated:
  * maximum concentration (Cmax)
  * time to achieve maximum concentration (Tmax)
  * absorption rate constant (ka)
  * elimination rate constant (kel)
  * half-life (t1/2)
  * area under the curve (AUC)
  Penetration into body fluids will be determined by comparing exposure (i.e. AUC, Cmax) ratios between the body fluid and plasma or comparison of concentrations in paired samples.

SECONDARY OUTCOMES:
Composite pharmacodynamic outcomes of understudied drugs in children | Data will be collected throughout the hospital or outpatient stay up to 90 days
  When applicable, Monte Carlo simulations will be performed to evaluate therapeutic target attainment rates (pharmacodynamics) in the population of interest. The final PK model and parameters estimated in the population PK analysis will be used to perform these simulations.
Biomarkers associated with understudied drugs in children | Data will be collected throughout the hospital or outpatient stay up to 90 days
  The dosing, sampling, and demographic information recorded on the electronic data collection forms will be merged with the bioanalytical information to create a biomarker dataset for each study drug. Biomarkers will be identified using metabolomics/proteomics and pharmacogenomics methodologies. Samples for biomarker analysis will be stored for future use in a PTN designated biorepository. Associations between biomarkers and drug exposure will be explored by visual inspection (i.e. scatter plots) and statistical comparisons as needed.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Hornik, PharmD, Principal Investigator — Duke University
Locations (52):
- United States (43):
  - Alaska Native Medical Center, Anchorage, Alaska
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California at San Diego Medical Center, La Jolla, California
  - Axis Clinical Trials, Los Angeles, California
  - University of California, Los Angeles Medical Center, Los Angeles, California
  - The Children's Hospital Colorado, Aurora, Colorado
  - Yale New Haven Children's Hospital, New Haven, Connecticut
  - Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Jacksonville Shands Medical Center, Jacksonville, Florida
  - Kapiolani Womens and Childrens Medical Center, Honolulu, Hawaii
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Fairway, Kansas
  - Children's Mercy Hospital and Clinics, Kansas City, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Science Center, New Orleans, Louisiana
  - Ochsner Baptist Clinical Trials Unit, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - University of Montana, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of New Mexico, Health Sciences Center, Albuquerque, New Mexico
  - UNC Hospital Neonatal-Perinatal Medicine, Chapel Hill, North Carolina
  - Duke University Medical Center (PICU / NICU), Durham, North Carolina
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Akron Children's Hospital, Cleveland, Ohio
  - Board of Regents of the University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of South Carolina, Columbia, South Carolina
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Children's Hospital, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - Manitoba Institute of Child Health, Winnipeg, Manitoba
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Hospital Sainte-Justine, Montreal, Quebec
- Israel (2):
  - Assaf Harofeh Medical Center, Zerifin, Tel Aviv
  - Schneider Children's Medical Center of Israel, Petah Tikva
- KK Women's and Children's Hospital Pte Ltd, Singapore, Singapore
- United Kingdom (2):
  - Southampton General Hospital, Southampton, Hampshire
  - Alder Hey Children's Hospital, Liverpool, Merseyside

IPD SHARING:
Plan to Share IPD: No
Completed study datasets (limited PHI) may be requested from https://pediatrictrials.org/data-sharing-opportunities Study data may be posted to the NICHD Data and Specimen Hub (DASH)

REFERENCES:
- [Result] Tremoulet A, Le J, Poindexter B, Sullivan JE, Laughon M, Delmore P, Salgado A, Ian-U Chong S, Melloni C, Gao J, Benjamin DK Jr, Capparelli EV, Cohen-Wolkowiez M; Administrative Core Committee of the Best Pharmaceuticals for Children Act-Pediatric Trials Network. Characterization of the population pharmacokinetics of ampicillin in neonates using an opportunistic study design. Antimicrob Agents Chemother. 2014 Jun;58(6):3013-20. doi: 10.1128/AAC.02374-13. Epub 2014 Mar 10. PMID 24614374
- [Result] Gonzalez D, Melloni C, Yogev R, Poindexter BB, Mendley SR, Delmore P, Sullivan JE, Autmizguine J, Lewandowski A, Harper B, Watt KM, Lewis KC, Capparelli EV, Benjamin DK Jr, Cohen-Wolkowiez M; Best Pharmaceuticals for Children Act - Pediatric Trials Network Administrative Core Committee. Use of opportunistic clinical data and a population pharmacokinetic model to support dosing of clindamycin for premature infants to adolescents. Clin Pharmacol Ther. 2014 Oct;96(4):429-37. doi: 10.1038/clpt.2014.134. Epub 2014 Jun 20. PMID 24949994
- [Result] Gonzalez D, Melloni C, Poindexter BB, Yogev R, Atz AM, Sullivan JE, Mendley SR, Delmore P, Delinsky A, Zimmerman K, Lewandowski A, Harper B, Lewis KC, Benjamin DK Jr, Cohen-Wolkowiez M; Best Pharmaceuticals for Children Act--Pediatric Trials Network Administrative Core Committee. Simultaneous determination of trimethoprim and sulfamethoxazole in dried plasma and urine spots. Bioanalysis. 2015;7(9):1137-49. doi: 10.4155/bio.15.38. PMID 26039810
- [Result] Hornik CP, Benjamin DK Jr, Smith PB, Pencina MJ, Tremoulet AH, Capparelli EV, Ericson JE, Clark RH, Cohen-Wolkowiez M; Best Pharmaceuticals for Children Act-Pediatric Trials Network. Electronic Health Records and Pharmacokinetic Modeling to Assess the Relationship between Ampicillin Exposure and Seizure Risk in Neonates. J Pediatr. 2016 Nov;178:125-129.e1. doi: 10.1016/j.jpeds.2016.07.011. Epub 2016 Aug 10. PMID 27522443
- [Result] Gonzalez D, Delmore P, Bloom BT, Cotten CM, Poindexter BB, McGowan E, Shattuck K, Bradford KK, Smith PB, Cohen-Wolkowiez M, Morris M, Yin W, Benjamin DK Jr, Laughon MM. Clindamycin Pharmacokinetics and Safety in Preterm and Term Infants. Antimicrob Agents Chemother. 2016 Apr 22;60(5):2888-94. doi: 10.1128/AAC.03086-15. Print 2016 May. PMID 26926644
- [Result] Autmizguine J, Melloni C, Hornik CP, Dallefeld S, Harper B, Yogev R, Sullivan JE, Atz AM, Al-Uzri A, Mendley S, Poindexter B, Mitchell J, Lewandowski A, Delmore P, Cohen-Wolkowiez M, Gonzalez D; the Pediatric Trials Network Steering Committee. Population Pharmacokinetics of Trimethoprim-Sulfamethoxazole in Infants and Children. Antimicrob Agents Chemother. 2017 Dec 21;62(1):e01813-17. doi: 10.1128/AAC.01813-17. Print 2018 Jan. PMID 29084742
- [Result] Le J, Poindexter B, Sullivan JE, Laughon M, Delmore P, Blackford M, Yogev R, James LP, Melloni C, Harper B, Mitchell J, Benjamin DK Jr, Boakye-Agyeman F, Cohen-Wolkowiez M. Comparative Analysis of Ampicillin Plasma and Dried Blood Spot Pharmacokinetics in Neonates. Ther Drug Monit. 2018 Feb;40(1):103-108. doi: 10.1097/FTD.0000000000000466. PMID 29271816
- [Result] Dallefeld SH, Atz AM, Yogev R, Sullivan JE, Al-Uzri A, Mendley SR, Laughon M, Hornik CP, Melloni C, Harper B, Lewandowski A, Mitchell J, Wu H, Green TP, Cohen-Wolkowiez M. A pharmacokinetic model for amiodarone in infants developed from an opportunistic sampling trial and published literature data. J Pharmacokinet Pharmacodyn. 2018 Jun;45(3):419-430. doi: 10.1007/s10928-018-9576-y. Epub 2018 Feb 12. PMID 29435949
- [Result] Hornik CP, Gonzalez D, van den Anker J, Atz AM, Yogev R, Poindexter BB, Ng KC, Delmore P, Harper BL, Melloni C, Lewandowski A, Gelber C, Cohen-Wolkowiez M, Lee JH; Pediatric Trial Network Steering Committee. Population Pharmacokinetics of Intramuscular and Intravenous Ketamine in Children. J Clin Pharmacol. 2018 Aug;58(8):1092-1104. doi: 10.1002/jcph.1116. Epub 2018 Apr 20. PMID 29677389
- [Result] Drolet BA, Boakye-Agyeman F, Harper B, Holland K, Lewandowski A, Stefanko N, Melloni C; Pediatric Trials Network Steering Committee (See Acknowledgments for a listing of committee members.). Systemic timolol exposure following topical application to infantile hemangiomas. J Am Acad Dermatol. 2020 Mar;82(3):733-736. doi: 10.1016/j.jaad.2019.02.029. Epub 2019 Feb 18. No abstract available. PMID 30790601
- [Result] Hornik CP, Yogev R, Mourani PM, Watt KM, Sullivan JE, Atz AM, Speicher D, Al-Uzri A, Adu-Darko M, Payne EH, Gelber CE, Lin S, Harper B, Melloni C, Cohen-Wolkowiez M, Gonzalez D; Best Pharmaceuticals for Children Act-Pediatric Trials Network Steering Committee. Population Pharmacokinetics of Milrinone in Infants, Children, and Adolescents. J Clin Pharmacol. 2019 Dec;59(12):1606-1619. doi: 10.1002/jcph.1499. Epub 2019 Jul 17. PMID 31317556
- [Result] Maharaj AR, Gonzalez D, Cohen-Wolkowiez M, Hornik CP, Edginton AN. Improving Pediatric Protein Binding Estimates: An Evaluation of alpha1-Acid Glycoprotein Maturation in Healthy and Infected Subjects. Clin Pharmacokinet. 2018 May;57(5):577-589. doi: 10.1007/s40262-017-0576-7. PMID 28779462
- [Result] Maharaj AR, Wu H, Zimmerman KO, Speicher DG, Sullivan JE, Watt K, Al-Uzri A, Payne EH, Erinjeri J, Lin S, Harper B, Melloni C, Hornik CP; Best Pharmaceuticals for Children Act - Pediatric Trials Network Steering Committee. Dosing of Continuous Fentanyl Infusions in Obese Children: A Population Pharmacokinetic Analysis. J Clin Pharmacol. 2020 May;60(5):636-647. doi: 10.1002/jcph.1562. Epub 2019 Dec 8. PMID 31814149
- [Result] Thompson EJ, Wu H, Melloni C, Balevic S, Sullivan JE, Laughon M, Clark KM, Kalra R, Mendley S, Payne EH, Erinjeri J, Gelber CE, Harper B, Cohen-Wolkowiez M, Hornik CP; Best Pharmaceuticals for Children Act - Pediatric Trials Network Steering Committee. Population Pharmacokinetics of Doxycycline in Children. Antimicrob Agents Chemother. 2019 Sep 9;63(12):e01508-19. doi: 10.1128/AAC.01508-19. Epub 2019 Sep 23. PMID 31548185
- [Result] Ge S, Mendley SR, Gerhart JG, Melloni C, Hornik CP, Sullivan JE, Atz A, Delmore P, Tremoulet A, Harper B, Payne E, Lin S, Erinjeri J, Cohen-Wolkowiez M, Gonzalez D; Best Pharmaceuticals for Children Act - Pediatric Trials Network Steering Committee. Population Pharmacokinetics of Metoclopramide in Infants, Children, and Adolescents. Clin Transl Sci. 2020 Nov;13(6):1189-1198. doi: 10.1111/cts.12803. Epub 2020 May 27. PMID 32324313
- [Result] Maharaj AR, Wu H, Zimmerman KO, Autmizguine J, Kalra R, Al-Uzri A, Sherwin CMT, Goldstein SL, Watt K, Erinjeri J, Payne EH, Cohen-Wolkowiez M, Hornik CP. Population pharmacokinetics of olanzapine in children. Br J Clin Pharmacol. 2021 Feb;87(2):542-554. doi: 10.1111/bcp.14414. Epub 2020 Jul 5. PMID 32497307
- [Result] Commander SJ, Wu H, Boakye-Agyeman F, Melloni C, Hornik CD, Zimmerman K, Al-Uzri A, Mendley SR, Harper B, Cohen-Wolkowiez M, Hornik CP; Best Pharmaceuticals for Children Act-Pediatric Trials Network Steering Committee. Pharmacokinetics of Hydrochlorothiazide in Children: A Potential Surrogate for Renal Secretion Maturation. J Clin Pharmacol. 2021 Mar;61(3):368-377. doi: 10.1002/jcph.1739. Epub 2020 Oct 7. PMID 33029806
- [Result] Wu YSS, Cohen-Wolkowiez M, Hornik CP, Gerhart JG, Autmizguine J, Cobbaert M, Gonzalez D; Best Pharmaceuticals for Children Act-Pediatric Trials Network Steering Committee. External Evaluation of Two Pediatric Population Pharmacokinetics Models of Oral Trimethoprim and Sulfamethoxazole. Antimicrob Agents Chemother. 2021 Jun 17;65(7):e0214920. doi: 10.1128/AAC.02149-20. Epub 2021 Jun 17. PMID 33903114
- [Result] Maharaj AR, Wu H, Zimmerman KO, Muller WJ, Sullivan JE, Sherwin CMT, Autmizguine J, Rathore MH, Hornik CD, Al-Uzri A, Payne EH, Benjamin DK Jr, Hornik CP; Best Pharmaceuticals for Children Act-Pediatric Trials Network Steering Committee. Pharmacokinetics of Ceftazidime in Children and Adolescents with Obesity. Paediatr Drugs. 2021 Sep;23(5):499-513. doi: 10.1007/s40272-021-00460-4. Epub 2021 Jul 23. PMID 34302290
- [Result] Gerhart JG, Carreno FO, Ford JL, Edginton AN, Perrin EM, Watt KM, Muller WJ, Atz AM, Al-Uzri A, Delmore P, Gonzalez D; Best Pharmaceuticals for Children Act-Pediatric Trials Network Steering Committee. Use of physiologically-based pharmacokinetic modeling to inform dosing of the opioid analgesics fentanyl and methadone in children with obesity. CPT Pharmacometrics Syst Pharmacol. 2022 Jun;11(6):778-791. doi: 10.1002/psp4.12793. Epub 2022 May 2. PMID 35491971
- [Result] Karatza E, Ganguly S, Hornik CD, Muller WJ, Al-Uzri A, James L, Balevic SJ, Gonzalez D. External Evaluation of Risperidone Population Pharmacokinetic Models Using Opportunistic Pediatric Data. Front Pharmacol. 2022 Mar 17;13:817276. doi: 10.3389/fphar.2022.817276. eCollection 2022. PMID 35370711
- [Result] Smith MJ, Gonzalez D, Goldman JL, Yogev R, Sullivan JE, Reed MD, Anand R, Martz K, Berezny K, Benjamin DK Jr, Smith PB, Cohen-Wolkowiez M, Watt K; Best Pharmaceuticals for Children Act-Pediatric Trials Network Steering Committee. Pharmacokinetics of Clindamycin in Obese and Nonobese Children. Antimicrob Agents Chemother. 2017 Mar 24;61(4):e02014-16. doi: 10.1128/AAC.02014-16. Print 2017 Apr. PMID 28137820
- [Derived] Hornik CP, Wu H, Edginton AN, Watt K, Cohen-Wolkowiez M, Gonzalez D. Development of a Pediatric Physiologically-Based Pharmacokinetic Model of Clindamycin Using Opportunistic Pharmacokinetic Data. Clin Pharmacokinet. 2017 Nov;56(11):1343-1353. doi: 10.1007/s40262-017-0525-5. PMID 28290120
- See also: Understudied Drugs Project Summary — https://pediatrictrials.org/pharmacokinetics-of-understudied-drugs-administered-to-children-per-standard-of-care-ptn-pops/